CLINICAL TRIAL: NCT06807021
Title: Post-operative Topical Administration of Fibrosis Inhibiting Compound FS2 in a Double- Blind, Randomized, Vehicle-controlled Study Evaluating the Safety and Mitigation of Cutaneous Scarring in Skin Graft and Donor Sites in Burn Patients
Brief Title: Post-Operative Use of FS2 to Mitigate Scarring in Burn Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Birch BioMed Inc (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B04-23-01-T0058
Record Dates: First submitted 2025-01-22; First posted 2025-02-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Burn Scar; Burn Wound
Keywords: Scar; Burn; skin graft; Kynurenic acid; FS2; Skin grafted wound; Donor Wound
MeSH Terms: conditions — Burns; Cicatrix | interventions — I-kappa B Kinase

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, vehicle-controlled, Randomized, Double-blinded
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Grafted wound (Experimental): The wound site (injury)
  Interventions: Drug: IP1 control cream (Vehicle base); Drug: IP2 - 0.5% w/w FS2
- Donor Skin Graft Harvest wound (Experimental): A Surgical wound
  Interventions: Drug: IP1 control cream (Vehicle base); Drug: IP2 - 0.5% w/w FS2

INTERVENTIONS:
Drug: IP1 control cream (Vehicle base) — Without FS2
Drug: IP2 - 0.5% w/w FS2 — FS2 in pharmaceutical compounding base

SUMMARY:
The goal of this study is to see how an ingredient called kynurenic acid (which we named "FS2") affects scar formation in people with burn injuries that need skin graft surgery. A cream with FS2 will be used on both the area where the skin graft was placed and the area where the skin was taken (donor site). The cream will be applied after the skin has healed. This study will help us understand if FS2 is safe and effective for mitigating skin scar formation in burn patients.

DETAILED DESCRIPTION:
For the first 90 days of the study, neither the patient nor the investigator will know which cream is being used: either the control cream (IP1) or the treatment cream (IP2), which contains 0.5% FS2. The assigned study product will be applied to the donor site and the skin graft site. After the first 90 days, all patients will use the FS2 cream for another 90 days in an open-label period where everyone knows they are receiving FS2.

The graft and donor sites will be photographed and assessed (POSAS and VSS), scored and recorded at the initial visit and again at every assessment visit thereafter.

An interim analysis will take place when about half of the participants (36 people) have finished their Day 90 visit. Based on the results, the study may continue as planned with the two-treatment, blinded design, or it may switch to an open-label format where all patients (those already in the study or newly enrolled) will use the FS2 cream.

Oversight - Human Subjects Protection Review section continued:

Site #02 (Edmonton) Approval Number: Pro00151882 Board Name: HREB - Biomedical Panel Board Affiliation: HREB - University of Alberta Board Contact Information: 780-492-8320 (Phone), vnadeau@ualberta.ca (Email)

ELIGIBILITY:
Inclusion Criteria:

1. Medically able and willing to consent to study requirements
2. Adult, male and female burn patients
3. Ages 18 to 60 years of age
4. Able to understand the study requirements and consent without a translator
5. Have a BMI between 15 and 35 kg/m2 (inclusive)
6. Have clinically acceptable results in the safety laboratory tests as deemed by the investigator
7. Have full thickness burn injury that requires partial thickness skin graft (meshed) for any location other than the face and genitalia
8. Meshed skin graft size is between 50 cm2 and 800 cm2
9. Maximum skin graft expansion ratio is 1:1.5
10. Able to apply the IPs as instructed, whether by the participants themselves or their accompanying caregivers

Exclusion Criteria:

1. Medically unable to consent to study requirements
2. Treatment site(s) (skin graft site) located on the face and genitalia
3. Treatment site(s) (skin graft site) take more than 14 days after the skin graft surgery to reach complete re-epithelization, based on the investigator's assessment
4. Expected to be medically unstable for the duration of the study period and an additional 1-month thereafter
5. Pregnant, or attempting to become pregnant
6. Subjects who had taken part in an interventional clinical trial within 3 months prior to admission to this trial or who are currently participating in a clinical trial, whether an investigational drug was used or not
7. Subjects who had any clinical evidence of severe ongoing or prolonged depression or mental illness within the last year
8. Subjects who smoke more than 20 cigarettes a day
9. Subjects who have a history of heavy drinking in the past month, defined as more than 14 drinks per week for men or more than 7 drinks per week for women
10. Subjects who have a history of substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention)
11. Subjects with severe inhalation injury requiring FiO2 >50%, renal failure requiring dialysis or hemodynamic instability requiring vasopressor therapy at the time of initiation of study treatment
12. Subjects who have scarring from previous interventions or evidence of thermal, electrical or radiation burn scars, tattoos, birthmarks or moles within 5 cm of the treatment sites
13. Subjects with a history of abnormal keloid scarring
14. Subjects with additional concurrent illnesses or conditions that may have interfered with wound healing like neoplastic, immune-mediated, or primary infectious disease (e.g. carcinoma, vasculitis, connective tissue disease, immune system disorders, uncontrolled HIV infection, rheumatoid arthritis, chronic renal impairment, significant hepatic impairment, inadequately or uncontrolled congestive heart failure or diabetes mellitus) or any clinically significant medical condition or history of any condition which may impair wound healing
15. Subjects with a skin disorder that is chronic or currently active and which the investigator considers will adversely affect the healing of acute wounds or will involve the areas to be examined in this trial (including psoriasis, dermatitis, eczema)
16. A history of radiotherapy to the study scar area
17. Subjects who have known sensitivities to any components of the IPs
18. Any other diagnosis, condition, physical or geographical limitation with the participant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Scar condition of the skin grafted wound on Day 90 as assessed by VSS | 90 days
  To evaluate the effect of 90-day FS2 cream use, compared to control, on clinician-assessed scar condition assessed by Vancouver Scar Scale (VSS) at the skin grafted wound (Study Arm 1)

SECONDARY OUTCOMES:
Scar condition of the donor skin graft harvest site on Day 90 as assessed by VSS | 90 days
  To evaluate the effect of 90-day FS2 cream use, compared to control, on clinician-assessed scar condition assessed by VSS at the donor skin graft harvest site (Study Arm 2)
Scar condition of the skin graft wound on Day 28 and Day 60 as assessed by VSS | Day 28 and Day 60
  To evaluate the effect of 28- and 60-day FS2 cream use, compared to control, on clinician-assessed scar condition assessed by VSS at: skin grafted wound (Study Arm 1)
Scar condition of the donor skin graft harvest site on Day 28 and Day 60 as assessed by VSS | Day 28 and Day 60
  To evaluate the effect of 28- and 60-day FS2 cream use, compared to control, on clinician-assessed scar condition assessed by VSS at: donor skin graft harvest site (Study Arm 2)
Scar condition of the skin grafted wound on Day 28, Day 60, and Day 90 as assessed by the Observer component of POSAS | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60- and 90-day FS2 cream use, compared to control, on clinician-assessed scar condition assessed by the Observer component of Patient and Observer Scar Assessment Scale (POSAS) at skin grafted wound (Study Arm 1)
Scar condition of the donor skin graft harvest site on Day 28, Day 60, and Day 90 as assessed by the Observer component of POSAS | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60- and 90-day FS2 cream use, compared to control, on clinician-assessed scar condition assessed by (POSAS) at: donor skin graft harvest site (Study Arm 2)
Scar condition of the skin grafted wound on Day 28, Day 60, and Day 90 as assessed by the Patient component of POSAS | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60- and 90-day FS2 cream use, compared to control, on patient-reported scar condition at: skin grafted wound (Study Arm 1)
Scar condition of the donor skin graft harvest site on Day 28, Day 60, and Day 90 as assessed by the Patient component of POSAS | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60- and 90-day FS2 cream use, compared to control, on patient-reported scar condition at: donor skin graft harvest site (Study Arm 2)
Scar condition of the skin grafted wound on Day 120 and Day 180 as assessed by the Observer component of POSAS | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on clinician-assessed scar condition at: skin grafted wound (Study Arm 1) - POSAS
Scar condition of the donor skin graft harvest site on Day 120 and Day 180 as assessed by the Observer component of POSAS | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on clinician-assessed scar condition at: donor skin graft harvest site (Study Arm 2) - POSAS
Scar condition of the skin grafted wound on Day 120 and Day 180 as assessed by VSS | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on clinician-assessed scar condition at: skin grafted wound (Study Arm 1) - VSS
Scar condition of the donor skin graft harvest site on Day 120 and Day 180 as assessed by VSS | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on clinician-assessed scar condition at: donor skin graft harvest site (Study Arm 2) - VSS
Scar condition of the skin grafted wound on Day 120 and Day 180 as assessed by the Patient component of POSAS | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on patient-reported scar condition at: skin grafted wound (Study Arm 1) -POSAS
Scar condition of the donor skin graft harvest site on Day 120 and Day 180 as assessed by the Patient component of POSAS | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on patient-reported scar condition at: donor skin graft harvest site (Study Arm 2) - POSAS
Scar condition of the skin grafted wound on Day 120 and Day 180 as assessed by the Observer component of POSAS | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on clinician-assessed scar condition at: skin grafted wound (Study Arm 1) - POSAS
Scar condition of the donor skin graft harvest site on Day 120 and Day 180 as assessed by the Observer component of POSAS | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on clinician-assessed scar condition at: donor skin graft harvest site (Study Arm 2) - POSAS
Scar condition of the skin grafted wound on Day 120 and Day 180 as assessed by VSS | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on clinician-assessed scar condition at: skin grafted wound (Study Arm 1) - VSS
Scar condition of the donor skin graft harvest site on Day 120 and Day 180 as assessed by VSS | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on clinician-assessed scar condition at: donor skin graft harvest site (Study Arm 2) - VSS
Scar condition of the skin grafted wound on Day 120 and Day 180 as assessed by the Patient component of POSAS | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on patient-reported scar condition at: skin grafted wound (Study Arm 1)
Scar condition of the donor skin graft harvest site on Day 120 and Day 180 as assessed by the Patient component of POSAS | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on patient-reported scar condition at: donor skin graft harvest site (Study Arm 2)
Quality of life on Day 28, Day 60, and Day 90 as assessed by the Burn Specific Health Scale-Brief (BSHS-B) | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60- and 90-day FS2 cream use, compared to control, on burn injury-related quality of life
Quality of life on Day 120 and Day 180 as assessed by BSHS-B | Day 120 and Day 180
  Quality of life on Day 120 and Day 180 as assessed by BSHS-B To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on burn injury-related quality of life in those randomized to control for the first 90 days of study
Quality of life on Day 120 and Day 180 as assessed by BSHS-B | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on burn injury-related quality of life in those randomized to FS2 cream for the first 90 days of study Quality of life on Day 120 and Day 180 as assessed by BSHS-B

OTHER OUTCOMES:
Scar size(cm2) at the skin grafted wound on Day 28, Day 60 and Day 90 as assessed by photographs | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60-, and 90-day FS2 cream use, compared to control, on wound scarring from: skin grafted wound (Study Arm 1)
Scar height(cm) at the skin grafted wound on Day 28, Day 60 and Day 90 as assessed by photographs | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60-, and 90-day FS2 cream use, compared to control, on wound scarring from: skin grafted wound (Study Arm 1)
Scar size(cm2) at the donor skin graft harvest site on Day 28, Day 60 and Day 90 as assessed by photographs | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60-, and 90-day FS2 cream use, compared to control, on wound scarring from: donor skin graft harvest site (Study Arm 2)
Scar height(cm) at the donor skin graft harvest site on Day 28, Day 60 and Day 90 as assessed by photographs | Day 28, Day 60 and Day 90
  To evaluate the effect of 28-, 60-, and 90-day FS2 cream use, compared to control, on wound scarring from: donor skin graft harvest site (Study Arm 2)
Scar size(cm2) at the skin grafted wound on Day 120 and Day 180 as assessed by photographs | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on wound scarring from: skin grafted wound (Study Arm 1)
Scar height(cm) at the skin grafted wound on Day 120 and Day 180 as assessed by photographs | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on wound scarring from: skin grafted wound (Study Arm 1)
Scar size(cm2)at the donor skin graft harvest site on Day 120 and Day 180 as assessed by photographs | Day 120 and Day 180
  To evaluate the effect of 120- and 180-day FS2 cream use on wound scarring from: donor skin graft harvest site (Study Arm 2)
Scar height(cm) at the donor skin graft harvest site on Day 120 and Day 180 as assessed by photographs | Day 120 and Day 180
  To evaluate the effect of 30- and 90-day FS2 cream use, starting 90 days after skin grafted wound's complete re-epithelization, on wound scarring from: donor skin graft harvest site (Study Arm 2)
To evaluate the Safety of FS2 Cream - Adverse events | Day 0, Day 28, Day 60, Day 90 and Day 180
  Report of Adverse Events
To evaluate the safety of FS2 cream - Whole Blood Hemoglobin (g/dl) | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Hematocrit (%) | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Red Blood Cell Count | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Red Cell distribution Width | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Mean corpuscular Volume | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Mean corpuscular Hemoglobin | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Mean corpuscular Hemoglobin Concentration | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - White Blood Cell Count and Differential | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Platelet Count | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - Mean Platelet Volume | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory Parameters - Hematology Parameters (Complete blood count)
To evaluate the safety of FS2 cream - AST | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety Laboratory parameters: Clinical Chemical Parameters
To evaluate the safety of FS2 cream - ALT | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety laboratory parameters: Clinical chemistry parameters:
To evaluate the safety of FS2 cream - GGT | Day 0, Day 28, Day 60, Day 90 and Day 180
  To evaluate the safety of FS2 cream Safety laboratory parameters: Clinical chemistry parameters.
To evaluate the safety of FS2 cream - Alkaline Phosphate | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety laboratory parameters: Clinical chemistry parameters
To evaluate the safety of FS2 cream - Creatinine | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety laboratory parameters Clinical chemistry parameters.
To evaluate the safety of FS2 cream - BUN | Day 0, Day 28, Day 60, Day 90 and Day 180
  To evaluate the safety of FS2 cream Safety laboratory parameters: Clinical chemistry parameters.
To evaluate the safety of FS2 cream - Bilirubin Total | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety laboratory parameters: Clinical chemistry parameters.
To evaluate the safety of FS2 cream - Bilirubin Direct | Day 0, Day 28, Day 60, Day 90 and Day 180
  Safety laboratory parameters: Clinical chemistry parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Camozzi, MD, PHD, Study Director — BirchBioMed Inc.
Locations (2):
- Canada (2):
  - University of Alberta, Division of Plastic Surgery, Edmonton, Alberta
  - Centre for Burn Research - Hamilton Health Sciences, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No